CLINICAL TRIAL: NCT00004697
Title: Randomized Study of the Use of Intravenous Choline Supplementation in Long Term Total Parenteral Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13360; UT-H-HSC-MS-97-018; BCM-FDR001118
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-03

CONDITIONS: Fatty Liver
Keywords: gastrointestinal disorders; hepatic steatosis; rare disease
MeSH Terms: conditions — Fatty Liver; Gastrointestinal Diseases; Rare Diseases | interventions — Choline

INTERVENTIONS:
Drug: choline chloride

SUMMARY:
OBJECTIVES:

I. Determine whether intravenous choline supplementation will reverse the hepatic steatosis and improve liver function in patients who receive long term total parenteral nutrition.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, double blind, placebo controlled study.

Patients receive either daily choline chloride in their total parenteral nutrition (TPN) solution or their usual TPN. The TPN is given intravenously over a 12 hour period beginning at approximately 9 PM nightly. Therapy continues for 24 weeks. Adjustments in the daily dose of choline provided may be required based on plasma free choline levels and patient tolerance. Additionally, all patients record the type and amount of their food intake on a daily basis.

Patients are followed every 2 weeks during the first 6 weeks, then every 4 weeks beginning with week 12 for the remainder of the 24 weeks, and then again at week 34.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Receiving nightly total parenteral nutrition (TPN) for greater than 70% of nutritional needs for a minimum of 8 weeks prior to study entry; Receiving no greater than 38 kcal/kg/day/ideal body weight; Receiving lipid emulsion as part of TPN regimen

Expected to require TPN for at least 34 weeks after study entry

Hepatic steatosis documented by prestudy CT scan

Consistent daily amount of intravenous amino acids, dextrose, or lipid received for 3 weeks prior to study entry

--Prior/Concurrent Therapy--

No concurrent cholinergic medications

--Patient Characteristics--

Hepatic: Albumin at least 3.5 g/dL; No hepatic failure; PT no greater than 2 times upper limit of normal

Renal: No renal failure requiring hemo- or peritoneal dialysis

Other: No AIDS; Not pregnant or nursing; Negative pregnancy test; Fertile patients must use effective contraception

Ages: 16 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 1997-11; Study Completion 1999-03

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lewis Buchman, Study Chair — University of Texas